CLINICAL TRIAL: NCT00018252
Title: The Effect of Exercise Training on Mental Stress-Induced Silent Ischemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized
Other Study IDs: AGCG-003-96F
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2001-06

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia | interventions — Exercise

INTERVENTIONS:
Behavioral: exercise

SUMMARY:
Coronary artery disease (CAD) remains the leading cause of death in the elderly. Silent myocardial ischemia (SI) is a manifestation of CAD in which there is a transient alteration in myocardial perfusion, function, and/or electrical activity not accompanied by chest pain. Mental and emotional stress, in particular hostility and anger are potent inducers of SI, Individuals with SI are at a 3-5 fold higher risk for the development of angina, myocardial infarction and death than subjects without SI.

DETAILED DESCRIPTION:
The hypothesis of this study is that older individuals with occult cad, mental stress/ emotional arousal (anger) increases sympathetic nervous system activity resulting in vasoconstriction thereby eliciting transient episodes of SI. Therefore an aerobic exercise intervention that reduces the response to anger/hostility and improves vascular compliance will decrease the ischemic burden in SI patients. The specific objectives are: To determine if non-smoking older individuals with exercise-induced SI have increased vasoreactivity (blood pressure, heart rate) responses to the laboratory presentation of mental stressors, decreased vascular compliance and brachial artery endothelial reactivity compared to matched non-ischemic controls; 2) To perform a randomized clinical trial that will examine the effects of 9 months of aerobic exercise training versus usual care on vasoreactivity, vascular compliance and ischemic burden on Holter monitor. Older individuals without a history of overt CAD will be recruited and evaluated for the presence of exercise-induced SI. Baseline cross-sectional comparisons of vasoreactivity and cardiovascular function will be performed between those with SI and non-ischemic controls. The individuals with SI will be enrolled in a randomized clinical trial of exercise vs usual care. Exercise treadmill testing with measurement of maximal aerobic capacity will be used to determine fitness. Vasoactivity will be quantified during a mental stress test with real time 2d echo imaging. Vascular function will be assessed using high frequency ultrasound measurements of flow-mediated brachial artery endothelial reactivity.

ELIGIBILITY:
Older individuals without a history of overt CAD.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 1997-04; Study Completion 2000-03

CONTACTS AND LOCATIONS:
Locations (1):
- VA Maryland Health Care System, Baltimore, Maryland, United States